CLINICAL TRIAL: NCT05957744
Title: Nutritional Risk Factors in Patients With Colorectal Cancer
Brief Title: Nutritional Risk Factors and Colorectal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Clinic Dr Dragisa Misovic-Dedinje (Other)
Responsible Party: Principal Investigator, Marina Boboš, Assistant Professor Dr., University Clinic Dr Dragisa Misovic-Dedinje
Other Study IDs: /2-2023
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Nutrition Related Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with colorectal cancer and malnutrition
  Interventions: Procedure: Colorectal surgery
- Group with colorectal cancer without malnutrition
  Interventions: Procedure: Colorectal surgery

INTERVENTIONS:
Procedure: Colorectal surgery — Right hemicolectomy, left colectomy, total colectomy, anterior resection

SUMMARY:
This observational study aims to learn about the relationship between the nutritional status of patients with colorectal cancer and clinical outcome after colorectal surgery.

The main question[s] it aims to answer are:

* which anthropometric, laboratory and specific parameters best define that patient is at nutritional risk
* will patients that are at nutritional risk stay longer in the hospital after surgery than those who are not at nutritional risk Patients will be preoperatively examined anthropometrically, radiologically and laboratoryally. Postoperatively, the course of their treatment will be monitored, as well as the monitoring of postoperative complications. A group of patients with and without malnutrition will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* First operation of this type

Exclusion Criteria:

* Urgent surgery
* Peritoneal carcinomatosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable carcinoma of the colon or rectum
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Center "Dr. Dragisa Misovic, Dedinje", Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No